CLINICAL TRIAL: NCT00439465
Title: Adoptive Cellular Immunotherapy Following Autologous Peripheral Blood Stem Cell Transplantation for Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: The Leukemia and Lymphoma Society (Other)
Responsible Party: Principal Investigator, Kenneth Meehan, Director, Bone Marrow Transplant Program, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D0717
Record Dates: First submitted 2007-02-21; First posted 2007-02-23 (Estimated); Results first posted 2019-03-26 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Myeloma; Transplant-eligible Patients
MeSH Terms: conditions — Neoplasms, Plasma Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ex-vivo expanded effector cells (Other): Infusing IL-2 and GM-CSF post-Hematopoietic Stem Cell Transplant (HSCT)
  Interventions: Biological: Ex-vivo expanded effector cells

INTERVENTIONS:
Biological: Ex-vivo expanded effector cells — This trial will test if the combination of infusing ex vivo expanded cytotoxic effector cells with IL-2 and GM-CSF post-transplant will accelerate immune reconstitution, resulting in an effector cell-versus-myeloma effect and, possibly, improved clinical outcomes.

SUMMARY:
The purpose of this study is to determine whether the administration of highly effective "killer" cells (cytotoxic T cells), along with Interleukin-2 (IL-2) and Recombinant Human Granulocyte Colony Stimulating Factor (GM-CSF) immediately following Autologous Peripheral Blood Stem Cell Transplantation (APBSCT) will enhance anti-tumor immune reconstitution and improve outcome of Multiple Myeloma patients.

The overall hypothesis of this proposal is that immediately following APBSCT the immune reconstitution is optimal to administer "killer" cells, combined with the administration of IL-2 and GM-CSF.

ELIGIBILITY:
Inclusion Criteria:

Multiple Myeloma:

* Patients must meet criteria for diagnosis of Multiple Myeloma.
* Patient must meet either criterion listed below:

  * Stage I, II, or III newly diagnosed multiple myeloma
  * Progressive or relapsed disease in partial response (PR) or complete response (CR)
  * Primary refractory disease.
  * Relapsed refractory disease.
  * Patients may have received a prior autologous transplant.
* The patients must have recovered from all serious and life threatening effects of previous treatment at the time of study entry (unless this abnormality is believed to be due to the underlying myeloma).
* The patient must have adequate bone marrow function, i.e. a total white blood cell count (WBC) of > 2,000/ul, a Hemoglobin (Hgb) of > 7 gm/dl, and a platelet count of > 50,000/ul, unless this abnormality is believed to be due to the underlying myeloma.
* The patient must have adequate liver function, i.e. bilirubin <2.0 mg/dl, aspartate aminotransferase (SGOT), alanine aminotransferase (SGPT) not greater than 2 times the upper normal limit (unless this abnormality is believed to be due to the underlying myeloma).
* The patient must have adequate renal function, i.e. serum creatinine < 3.0 mg/dl, and/or creatinine clearance >50 ml/min. This eligibility criterion is excluded if renal insufficiency is believed to be secondary to myeloma.
* Age >18 years and < 75 years old
* The patient must have a Karnofsky status > 80%
* Patients must have a life expectancy of at least 12 weeks
* Left ventricular ejection fraction of > 45% by radionuclide scan or echocardiography
* Pulmonary function tests: forced vital capacity, Diffusing capacity of the lungs for carbon monoxide (DLCO) and expiratory volume in one second (FEV1) must be > 50% of predicted
* No significant co-morbid medical or psychiatric illness which would significantly compromise the patient's clinical care and chances of survival.
* Informed written consent must be obtained. Patients must be able to give informed consent as a prerequisite to this procedure. The Informed Consent form will become part of his/her permanent record and a copy will be given to the patient

Exclusion Criteria:

* Medical, social, or psychological factors which would prevent the patient from receiving or cooperating with the full course of therapy.
* Evidence on physical exam, lumbar puncture, computed tomography (CT), or magnetic resonance imaging (MRI) scan of central nervous system (CNS) involvement with malignancy
* Any clinically significant cardiac disease (angina, myocardial infarction, congestive heart failure, ventricular arrhythmias requiring therapy) or clinically significant obstructive/restrictive pulmonary disease
* Serology positive for human immunodeficiency virus (HIV) or human T-lymphotropic virus (HTLVI)
* Active hepatitis B or C
* History of seizures
* Concurrent or expected need for therapy with corticosteroids
* Active connective tissue disease
* Current "clinically significant" pleural effusion, pericardial effusion, or ascites
* Positive pregnancy test or presence of lactation
* Collection of fewer than 1 x 106 cluster of differentiation 34 positive (CD34+) cells/kg (peripheral blood stem cells). If the apheresis collection is inadequate based on this criteria, the patient will be removed from protocol and a marrow harvest may be performed
* A history of a second malignancy (other then squamous cell/ basal cell carcinoma of the skin or cervical dysplasia) must be reviewed by the Principal Investigator, before inclusion or exclusion in the study. Based upon the PI's review, this patient may be eligible (i.e., distant past history of a malignancy)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-01; Primary Completion 2012-10-15 (Actual); Study Completion 2012-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Meehan, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ex-vivo Expanded Effector Cells: Infusing Interleukin-2 (IL-2) and Recombinant Human Granulocyte Colony Stimulating Factor (GM-CSF)post-Hematopoietic stem cell transplant (HSCT)
  Ex-vivo expanded effector cells: This trial will test if the combination of infusing ex vivo expanded cytotoxic effector cells with IL-2 and GM-CSF post-transplant will accelerate immune reconstitution, resulting in an effector cell-versus-myeloma effect and, possibly, improved clinical outcomes.
Period: Overall Study
Arm/Group | Ex-vivo Expanded Effector Cells
Started | 23
Completed | 19
Not Completed | 4

BASELINE CHARACTERISTICS:
Groups:
- Ex-vivo Expanded Effector Cells: Infusing IL-2 and GM-CSF post-HCST
  Ex-vivo expanded effector cells: This trial will test if the combination of infusing ex vivo expanded cytotoxic effector cells with IL-2 and GM-CSF post-transplant will accelerate immune reconstitution, resulting in an effector cell-versus-myeloma effect and, possibly, improved clinical outcomes.
Arm/Group | Ex-vivo Expanded Effector Cells
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 6
Age, Continuous [Median (Full Range); unit: Years] | 60 [42 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events in All Subjects
Description: To establish the safety (toxicity) of myeloma patients treated with high dose melphalan, autologous peripheral blood stem cell transplantation (APBSCT) & adoptive transfer of cytotoxic effector cells with Interleukin-2 (IL-2) and Recombinant Human Granulocyte Colony Stimulating Factor (GM-CSF).
Time Frame: From initiation of treatment on protocol until Day 100
Measure: Count of Participants; unit: Participants
Groups:
- Ex-vivo Expanded Effector Cells: Infusing IL-2 and GM-CSF post-Hematopoietic Stem-Cell Transplant (HSCT) Ex-vivo expanded effector cells: This trial will test if the combination of infusing ex vivo expanded cytotoxic effector cells with IL-2 and GM-CSF post-transplant will accelerate immune reconstitution, resulting in an effector cell-versus-myeloma effect and, possibly, improved clinical outcomes.
Arm/Group | Ex-vivo Expanded Effector Cells
Number analyzed (Participants) | 23
Participants | 11

2. Secondary Outcome: Count of Participants With Increased CD3+CD8+, CD8+ and CD56+ Concentrations Between Day 15 Post-Transplant and Days 21 to 28 Post-transplant
Description: To demonstrate that the effector cell infusions result in a clinical effect, phenotypic analyses of blood samples using flow cytometry will be performed prior to, and after each infusion, focusing on the CD8 + populations (CD3+CD8+, CD8+CD56+). As a complement to flow cytometry, the following assays will be used to identify cell subset precursor frequencies, subset proliferation, and cytokine production:
  * Dye Dilution Proliferation Assay (DDPA) 36 - Evaluation of CD8+ T Cell Precursors
  * ELISPOT-Quantifying cytokine producing T cells:
Time Frame: Day 15 post-transplant and between days 21 to 28 post-transplant
Population: Sixteen out of nineteen subject samples were analyzed. Three subject's samples were not available for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Ex-vivo Expanded Effector Cells
Number analyzed (Participants) | 16
Participants
  Day 15: Increase | 7
  Day 15: No Increase | 9
  Days 21-28: Increase | 7
  Days 21-28: No Increase | 9

3. Secondary Outcome: Time to Recovery of Absolute Neutrophil Count
Description: To establish the time to engraftment of myeloma patients treated with high dose melphalan, APBSCT& adoptive transfer of cytotoxic effector cells with IL-2 and GM-CSF.
Time Frame: From initiation of treatment on protocol until Day 100
Measure: Median (Full Range); unit: Days
Arm/Group | Ex-vivo Expanded Effector Cells
Number analyzed (Participants) | 19
Days | 13 [12 to 16]

4. Secondary Outcome: Time to Recovery of Platelet Count
Description: as for outcome 3
Time Frame: From initiation of treatment on protocol until Day 100
Measure: Median (Full Range); unit: days
Arm/Group | Ex-vivo Expanded Effector Cells
Number analyzed (Participants) | 19
days | 16 [10 to 26]

5. Secondary Outcome: Assessment of Disease Response to Treatment
Description: To establish the disease response of myeloma patients treated with high dose melphalan, APBSCT& adoptive transfer of cytotoxic effector cells with IL-2 and GM-CSF.
Time Frame: From initiation of treatment on protocol until Day 100
Measure: Count of Participants; unit: Participants
Arm/Group | Ex-vivo Expanded Effector Cells
Number analyzed (Participants) | 19
Participants
  Complete Response | 12
  Very Good Partial Response | 5
  Partial Response | 1
  Progressive disease | 1

6. Secondary Outcome: Number of Participants With Increased Expression of DAP10 and NKG2D on the CD8 Cell Population
Description: * Isolate CD3+CD8+ and CD8+CD56+ from patients' blood following transplant.
  * Identify NKG2D and DAP10 expression.
  * Determine the mechanism of tumor cell killing and the relationship to NKG2D or DAP 10 expression.
  After isolating CD8+ cells from patient's blood samples using the AutoMACS, we will evaluate the expression of NKG2D and DAP10 on all CD8+ cells (CD3+CD8+ and CD8+CD56+cells) pre-transplant (Baseline) and following the third and fourth cellular infusions using phenotypic analysis. We postulate the increased expression of both DAP10 and NKG2D on the CD8 population immediately following APSCT and effector cell infusions when compared to baseline.
Time Frame: Pre-transplant and following the third and fourth cellular infusions
Population: Sixteen out of nineteen participants samples were analyzed. Three participants' samples were not available for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Ex-vivo Expanded Effector Cells
Number analyzed (Participants) | 16
Participants
  Increased abs. NKG2D+CD3+CD8 Tcells | 12
  Increased abs. NKG2D+CD3-CD56+ T cells | 12

7. Secondary Outcome: Determine the Methods of Tumor Cell Killing of the in Vivo CD8+ Cells: Cytotoxicity Assays, Blocking Experiments, Analysis of T-cell Receptor (TCR)
Description: We will isolate the CD8+ populations (CD3+CD8+, CD8+CD56+) using the Auto MACS (Miltenyi) and then identify the mechanisms of tumor cell killing by the CD8+ cells obtained pre-transplant (Baseline) and following the third and fourth cellular infusions. We will examine mechanisms of tumor cell killing through NKG2D receptor, major histocompatibility complex (MHC) Class I molecules or through the T cell receptor. We postulate the CD8+ cells obtained from patient's blood will kill tumor cells both via MHC Class I and through the NKG2D receptor.
Time Frame: Pre-transplant and following the third and fourth cellular infusions.
Population: Autologous myeloma cells were isolated for only 4 study participants. There is no information on the remaining participant provided.
Measure: Count of Participants; unit: Participants
Arm/Group | Ex-vivo Expanded Effector Cells
Number analyzed (Participants) | 5
Participants
  Autologous Myeloma Cells: number analyzed (Participants) | 4
  Autologous Myeloma Cells: Increased tumor lysis | 4
  Autologous Myeloma Cells: Failure of tumor lysis | 0
  Peripheral blood mononuclear cells: Increased tumor lysis | 5
  Peripheral blood mononuclear cells: Failure of tumor lysis | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the start of treatment until 100 days post-treatment for all subjects. Total time of adverse event collection for the study was January 2007 through March 2010
Arm/Group | Ex-vivo Expanded Effector Cells
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 11/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ex-vivo Expanded Effector Cells (N=23)
Moderate infection (Infections and infestations) | 3
Severe infection (Infections and infestations) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Increased liver function tests (Hepatobiliary disorders) | 2
anorexia (Metabolism and nutrition disorders) | 3
Mucositis - oral (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Fever (General disorders) | 2
Tachycardia (Cardiac disorders) | 2
Hypotension (Cardiac disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes